CLINICAL TRIAL: NCT01749059
Title: The Impact of Implementing a Universal Newborn Screening for Critical Congenital Heart Disease
Acronym: CCHD
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-003-11
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Congenital Heart Defect

SUMMARY:
The purpose of this study is to evaluate the impact of implementing a universal pulse oximeter screening as a way to detect critical congenital heart disease in otherwise well-appearing newborns.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of informed consent and authorization.
2. Full term and late preterm newborns (EGA 35-44 weeks)
3. On room air
4. Neonates known to have a congenital heart defect at the time of screening, e.g., antenatal diagnosis or diagnosis within the first 24 hours after birth
5. Parents agree to follow-up contact post discharge

Exclusion Criteria:

1. On supplemental oxygen
2. Admitted to the Neonatal Intensive Care Unit
3. Parents do not agree to follow-up
4. Greater than 30 days of age

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates known to have a congenital heart defect at the time of screening.
Sampling Method: Non-Probability Sample
Enrollment: 6147 (Actual)
Dates: Start 2012-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
True Positive Rate | One year follow-up
  The numbers of subjects who have a positive pulse oximetry screening test and who in follow-up evaluation are found to have CCHD.
False Positive Rate | One year follow-up
  The numbers of subjects who have a positive pulse oximetry screening test and who in follow-up evaluation are found to have normal hearts.
True Negative Rate | One year follow-up
  The number of subjects who have a negative pulse oximetry screening test and who in follow-up evaluation are found to have normal hearts.
False Negative Rate | One year follow-up
  The number of subjects who have a negative pulse oximetry screening test and who in follow-up evaluation are found to have heart defects.

CONTACTS AND LOCATIONS:
Overall Officials: Reese H Clark, MD, Principal Investigator — Pediatrix
Locations (1):
- Capital Health Regional Medical Center - Pediatrix Medical Group, Trenton, New Jersey, United States